CLINICAL TRIAL: NCT06309602
Title: Investigation of a Free Water Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Emily Main, MS, CCC-SLP, Principal Investigator, Poudre Valley Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0465
Record Dates: First submitted 2023-11-02; First posted 2024-03-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Oropharyngeal Dysphagia
Keywords: stroke; trauma
MeSH Terms: conditions — Deglutition Disorders; Stroke; Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control / Standard Care (Other): Standard care provided for patients with orders for thickened liquids.
  Interventions: Other: Control / Standard Care
- Free Water Protocol (Experimental): Standard care provided for patients with orders for thickened liquids. Additionally, participant will be allowed to have plain, un-thickened water after the following have taken place: 1) Wait 30 minutes after meal or medication administration; 2) Complete oral care according to instructions posted at bedside.
  Interventions: Other: Free Water Protocol

INTERVENTIONS:
Other: Free Water Protocol — Intake of plain, un-thickened water is allowed even when a patient has orders for thickened liquids. Risks of pulmonary complications are decreased with use of a strict oral care regimen and timed intake of water related to meals. Patient satisfaction and comfort is increased with ingestion of plain water.
  Arms: Free Water Protocol
Other: Control / Standard Care — Standard care will be given to patients with orders for thickened liquids. This will include oral care twice a day and implementation of swallowing strategies and precautions as prescribed by the treating speech-language pathologist. Only fluids thickened to the recommended viscosity will be available to the patient.
  Arms: Control / Standard Care

SUMMARY:
Hypothesis: Use of a Free Water Protocol (FWP) will improve patient satisfaction scores (Dysphagia Handicap Index), will not increase the risk of aspiration pneumonia/pneumonitis, and will result in improved oral hygiene (as assessed by the Oral Assessment Guide). Aim: To demonstrate that improvement in patient satisfaction and quality of life scores outweighs the potential risks of aspiration of plain water in an acute care setting; to qualitatively assess the implementation of a Free Water Protocol from the viewpoints of the patient and family/caregivers; to quantify changes in oral hygiene practices for individuals on the Free Water Protocol.

DETAILED DESCRIPTION:
Individuals who have difficulty swallowing thin liquids are commonly restricted from ingesting plain water and prescribed a thickened liquid only diet to prevent choking hazards and aspiration pneumonia. These thickened liquids are intended to reduce aspiration of oral secretions carrying respiratory pathogens, the primary cause of aspiration pneumonia. This restriction from plain water (also known as thin water) can result in lowered patient satisfaction in addition to dissatisfaction with the texture and taste of thickened liquids. However, prior research from inpatient rehabilitation settings has demonstrated that plain water can be given to patients who otherwise require thickened liquids to prevent aspiration pneumonia. If patients prescribed a thickened liquid diet are allowed access to plain water, then hydration status may improve along with increased patient satisfaction.

This Free Water Protocol (FWP) differs from a thickened-liquids-only protocol in three ways: 1) allowing individuals access to plain, un-thickened water; 2) purposefully providing oral care prior to access of plain water; and 3) not allowing plain water until 30 minutes after meal completion and oral care has been completed with the intent to reduce the risk of pulmonary complications. Although many institutions have adapted and implemented an FWP, only 10 studies have measured pulmonary complications of an FWP. Among those, other outcomes are reported inconsistently with varying methodologies (e.g., fluid intake, hydration status, occurrences of urinary tract infection, satisfaction measures). More research is needed to demonstrate the benefits of allowing free water over the risk of potential pulmonary complications, especially in an acute care setting.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis or trauma patients being cared for by Trauma & Acute Care Surgery (TACS) providers
* Current orders for restricted or thickened liquids
* Ability to control their own airway (i.e. airway adjuncts not needed)

Exclusion Criteria:

* Individuals who are medically fragile, as determined by treating physician, to include diagnosis of sepsis, need for vasopressors, or high oxygenation needs (requiring high-flow nasal cannula, Airvo, or oximask)
* Individuals who refuse oral care, have any decayed teeth or dental disease, or have a documented active oral infection
* Individuals with an advanced progressive neurological condition, active head/neck cancer, or those who are immunosuppressed
* Individuals who are on bed-rest orders
* Individuals who are lethargic or sedated
* Individuals with suspected pre-hospital aspiration event and/or aspiration pneumonitis
* Individuals with a fever of unknown origin
* Individuals with a history of recurrent aspiration pneumonia/pneumonitis
* Individuals whose primary language is one that the questionnaires are not available in a validated format

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Handicap Index | Through study completion, an average of 5 days
  Quality of life survey
Oral Assessment Guide | Through study completion, an average of 5 days
  8-point visual assessment of oral hygiene
Qualitative data | Through study completion, an average of 5 days
  Open-ended question to provide a narrative of patient impressions and satisfaction regarding eating and drinking

SECONDARY OUTCOMES:
Adverse events: Aspiration pneumonia/pneumonitis | Through study completion, an average of 5 days
  Aspiration pneumonia/pneumonitis diagnosed by the treating provider or by the following criteria: The presence of a new or evolving infiltrate on chest x-ray while meeting the following criteria: temperature greater than 38.2˚C, leukocytosis greater than 12,000 cells/mm3, and presence of purulent sputum or endotracheal aspirate)
Liquid intake | Through study completion, an average of 5 days
  Oral liquid volume consumed in 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States